CLINICAL TRIAL: NCT00120328
Title: ASCEND - A Randomised, Double Blind, Placebo Controlled, Parallel Group Study to Assess the Effect of the Endothelin Receptor Antagonist Avosentan on Time to Doubling of Serum Creatinine, End Stage Renal Disease or Death in Patients With Type 2 Diabetes Mellitus and Diabetic Nephropathy
Brief Title: To Determine the Effects of Avosentan on Doubling of Serum Creatinine, End Stage Renal Disease and Death in Diabetic Nephropathy
Status: Terminated | Phase: Phase 3 | Type: Interventional
Sponsor: Speedel Pharma Ltd. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: SPP301CRD15; 2005-000604-14
Record Dates: First submitted 2005-06-30; First posted 2005-07-15 (Estimated); Last update posted 2007-10-05 (Estimated); Status verified 2007-10

CONDITIONS: Diabetic Nephropathy
Keywords: serum creatinine; end stage renal disease; cardiovascular mortality; cardiovascular morbidity; non-cardiovascular mortality; non-cardiovascular morbidity
MeSH Terms: conditions — Diabetic Nephropathies; Kidney Failure, Chronic | interventions — Avosentan

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: SPP301

SUMMARY:
The purpose of this study is to determine whether avosentan (SPP301) is effective in decreasing morbidity and mortality in patients with diabetic nephropathy.

DETAILED DESCRIPTION:
Diabetic nephropathy has become the leading cause of end stage renal disease (ESRD) in the western world, accounting for approximately 40% of new cases in the US, and up to 20 to 30% in Europe.

Current treatments for diabetic nephropathy usually try to deal with the underlying diabetes or they aim to reduce cardiovascular risk factors such as hypertension, hyperglycemia, smoking and dyslipidemia. A few recently approved drugs such as irbesartan and losartan (for type 2 diabetic nephropathy) have a renoprotective activity beyond their antihypertensive effect. However, morbidity and mortality rates remain high.

Avosentan may have a positive effect on reducing the amount of protein lost in the urine and if this is the case it will help treat patients with diabetic nephropathy.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients between 21 and 80 years of age, inclusive
* Patients with type 2 diabetes mellitus diagnosed for at least 3 years and receiving oral anti-diabetic treatment and/or insulin
* Female patients will either be:

  * Post menopausal for >= 2 years;
  * Surgically sterile;
  * Or, if sexually active and of childbearing potential, using double contraception, with at least one method being barrier contraception. Women of childbearing potential (defined as those who are not surgically sterile, have not had a hysterectomy or are not 2 years' post-menopausal) must have a negative pregnancy test at screening and at randomisation. Pregnancy tests will be repeated monthly during the study
* Proteinuria defined as ACR >= 35mg/mmol
* Male patients with serum creatinine between 1.3 and 3.0 mg/dL
* Female patients with serum creatinine between 1.2 and 3.0 mg/dL
* On standard treatment for diabetic nephropathy (such as ACE inhibitors, ARBs or the combination thereof) for at least 6 months before screening. Patients who are intolerant to ACE inhibitors or ARBs will be allowed to enter the study
* Able to provide written informed consent prior to study participation

Exclusion Criteria:

* Patients with type 1 diabetes mellitus
* Patients with proteinuria of non-diabetic origin
* Patients with a renal transplant
* Patients who have undergone nephrectomy
* Patients with an estimated GFR <= 15 mL/min
* Patients with blood pressure >= 160/100 mmHg with or without antihypertensive medication
* Patients with glycosylated haemoglobin (HbA1c) > 12%
* Patients with normal sinus rhythm who do not have a pacemaker, are not taking antiarrhythmic drugs and do not have complete bundle branch block, but who have absolute QT or QTc >500 msec
* Patients with recent (60 days) percutaneous transluminal coronary angioplasty (PTCA), percutaneous coronary intervention (PCI), coronary artery bypass grafting (CABG), or any other major surgical intervention
* Patients with recent (60 days) acute myocardial infarction, unstable angina, stroke or transient ischaemic attack
* Patients with CHF New York Heart Association grade III or IV
* Patients with life-threatening arrhythmias including those at high risk for QT/QTc prolongation such as a family history of Long QT Syndrome, severe hypokalaemia, etc.
* Patients who are positive for hepatitis B surface antigen or hepatitis C antibody at Visit 1 (screening) and who have abnormal liver function (specifically ALAT/ASAT >1 x ULN)
* Patients who have been treated with an endothelin receptor antagonist in the 3 months prior to screening
* Patients being treated with spironolactone or eplerenone at entry into the study
* Pregnant or lactating women
* Patients with a neoplasm who are deemed to live < 12 months
* Patients with history of alcohol and/or drug abuse
* Patients with a known history of a major psychiatric condition that would interfere with the conduct of the trial
* Patients with active endocarditis and/or pericarditis
* Patients allergic to avosentan or any other endothelin receptor antagonist
* Patients who participated in another clinical study or who have donated blood within 60 days of being randomised to this study.

Ages: 21 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2364
Dates: Start 2005-07; Study Completion 2007-02 (Actual)

PRIMARY OUTCOMES:
To determine the effect of each dose of avosentan on time to doubling of serum creatinine, end stage renal disease (ESRD) or death when administered on top of standard treatment in subjects with type 2 diabetes mellitus and diabetic nephropathy.

SECONDARY OUTCOMES:
To determine the effect of each dose of avosentan on: cardiovascular mortality
non-cardiovascular mortality
coronary or peripheral vascular revascularisations including amputations (except where due to trauma)
non-fatal acute myocardial infarction
stroke
congestive heart failure
unstable angina

CONTACTS AND LOCATIONS:
Overall Officials: Jessica Mann, MD, PhD, Study Director — Speedel Pharma Ltd.
Locations (1):
- Dr. Mark Warren, Greenville, North Carolina, United States